CLINICAL TRIAL: NCT00320203
Title: A Study of the Safety and IOP-Lowering Efficacy of Anecortave Acetate in Patients With Open-Angle Glaucoma
Brief Title: Anecortave Acetate in Patients With Open-angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-04-62
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2008-02

CONDITIONS: Open-angle Glaucoma
Keywords: open-angle; glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — anecortave acetate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Anecortave Acetate 3 mg Depot (Experimental): Single injection, anterior juxtascleral depot (AJD)
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 6 mg/mL
- Anecortave Acetate 15 mg Depot (Experimental): Single injection, anterior juxtascleral depot (AJD)
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 30 mg/mL
- Anecortave Acetate 30 mg Depot (Experimental): Single injection, anterior juxtascleral depot (AJD)
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 60 mg/mL
- Anecortave Acetate Vehicle (Other): Single injection, anterior juxtascleral depot (AJD)
  Interventions: Other: Anecortave Acetate Vehicle

INTERVENTIONS:
Drug: Anecortave Acetate Sterile Suspension, 6 mg/mL — Single injection, anterior juxtascleral depot (AJD)
  Arms: Anecortave Acetate 3 mg Depot
Drug: Anecortave Acetate Sterile Suspension, 30 mg/mL — Single injection, anterior juxtascleral depot (AJD)
  Arms: Anecortave Acetate 15 mg Depot
Drug: Anecortave Acetate Sterile Suspension, 60 mg/mL — Single injection, anterior juxtascleral depot (AJD)
  Arms: Anecortave Acetate 30 mg Depot
Other: Anecortave Acetate Vehicle — Single injection, anterior juxtascleral depot (AJD)
  Arms: Anecortave Acetate Vehicle

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and duration of effect of a single administration of Anecortave Acetate Depot for treatment of elevated intraocular pressure (IOP) in patients with open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with open-angle glaucoma.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patients with open-angle glaucoma with a pseudoexfoliation or pigment dispersion component.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2006-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Mean change in intraocular pressure at 9 am from baseline | Weeks 2 and 6, Months 2, 3, 4, 5, 6, 7.5, 9, 10.5, and 12

SECONDARY OUTCOMES:
Time to treatment failure | At time point

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Landry, Study Director — Alcon Research